CLINICAL TRIAL: NCT02448420
Title: A Phase II Trial of Palbociclib in Combination With Trastuzumab and Endocrine Therapy in Patients With Previously-treated Locally Advanced or Metastatic HER2-positive Breast Cancer (PATRICIA II)
Brief Title: Study of Palbociclib and Trastuzumab With Endocrine Therapy in HER2-positive Metastatic Breast Cancer
Acronym: PATRICIA II
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: SOLTI Breast Cancer Research Group (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SOLTI-1303; 2014-005006-38 (EudraCT Number)
Record Dates: First submitted 2015-05-08; First posted 2015-05-19 (Estimated); Last update posted 2024-04-18 (Actual); Status verified 2024-04

CONDITIONS: Metastatic Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — palbociclib; Trastuzumab; Drug Therapy; Immunoconjugates; Ado-Trastuzumab Emtansine

STUDY DESIGN:
Intervention Model Description: When the recruitment cohorts C begins, the recruitment in cohorts A and B will be closed.
Oversight: Data Monitoring Committee: Yes

ARMS (5):
- Arm A: HER2-positive/Hormone receptor-negative (Recruitment Closed) (Experimental): Patients with hormone receptor-negative, HER2 positive breast cancer, who received trastuzumab + palbociclib.
  Palbociclib: oral, 200 mg/day for 2 weeks, followed by 1 week off. Trastuzumab: intravenous trastuzumab loading dose of 8mg/kg followed by 6 mg/kg once every 3 weeks; or subcutaneous trastuzumab 600mg every 3 weeks.
  Interventions: Drug: Palbociclib; Drug: Trastuzumab
- Arm B1: HER2+/Hormone receptor-positive (Recruitment Closed) (Experimental): Patients with hormone receptor-positive, HER2 positive breast cancer, who received trastuzumab + palbociclib.
  Palbociclib: oral, 200 mg/day for 2 weeks, followed by 1 week off. Trastuzumab: intravenous trastuzumab loading dose of 8mg/kg followed by 6 mg/kg once every 3 weeks; or subcutaneous trastuzumab 600mg every 3 weeks.
  Interventions: Drug: Palbociclib; Drug: Trastuzumab
- Arm B2:HER+/HR+: trastuzumab + palbociclib +letrozole (Recruitment Closed) (Experimental): Patients with hormone receptor-positive, HER2 positive breast cancer, who received trastuzumab + palbociclib + letrozole Palbociclib: oral, 200 mg/day for 2 weeks, followed by 1 week off. Trastuzumab: intravenous trastuzumab loading dose of 8mg/kg followed by 6 mg/kg once every 3 weeks; or subcutaneous trastuzumab 600mg every 3 weeks.
  Letrozole: daily oral dose of 2.5 mg.
  Interventions: Drug: Palbociclib; Drug: Trastuzumab; Drug: Endocrine therapy
- Arm C1: Palbociclib, trastuzumab and endocrine therapy (Experimental): HR-positive, HER2 positive, Luminal intrinsic subtype determined by PAM50 who will receive trastuzumab + palbociclib + endocrine therapy
  Trastuzumab: intravenous trastuzumab loading dose of 8mg/kg followed by 6 mg/kg once every 3 weeks; or subcutaneous trastuzumab 600mg every 3 weeks.
  Palbociclib: oral, 125 mg/d for 3 weeks, followed by one week off, in 4-week cycles.
  Endocrine therapy: either an Aromatase Inhibitor, Fulvestrant, or Tamoxifen.
  Interventions: Drug: Palbociclib; Drug: Trastuzumab; Drug: Endocrine therapy
- Arm C2: Treatment based of physician's choice (Active Comparator): HR-positive, HER2 positive, Luminal intrinsic subtype determined by PAM50 who will receive treatment based on physician's choice from the following options: TDM1 or chemotherapy (gemcitabine, vinorelbine, capecitabine, eribulin or a taxane) in combination with trastuzumab or endocrine therapy (Aromatase Inhibitor, Fulvestrant or Tamoxifen) in combination with trastuzumab.
  Interventions: Drug: Trastuzumab; Drug: Endocrine therapy; Drug: Chemotherapy; Drug: Antibody-Drug Conjugates

INTERVENTIONS:
Drug: Palbociclib — Cohort A, B1 y B2: Palbociclib oral dose of 200 mg/day for 2 weeks, followed by 1 week off.
  Cohort C1: Palbociclib oral dose 125 mg/d for 3 weeks, followed by one week off, in 4-week cycles.
  Other Names: Ibrance
  Arms: Arm A: HER2-positive/Hormone receptor-negative (Recruitment Closed); Arm B1: HER2+/Hormone receptor-positive (Recruitment Closed); Arm B2:HER+/HR+: trastuzumab + palbociclib +letrozole (Recruitment Closed); Arm C1: Palbociclib, trastuzumab and endocrine therapy
Drug: Trastuzumab — Loading dose of 8mg/kg intravenous (iv) followed by 6 mg/kg once every 3 weeks; or subcutaneous trastuzumab 600mg every 3 weeks.
  Other Names: Herceptin
Drug: Endocrine therapy — Non-steroidal AIs (anastrozole, letrozole); steroidal AI (exemestane); Fulvestrant or Tamoxifen
  Other Names: ET
  Arms: Arm B2:HER+/HR+: trastuzumab + palbociclib +letrozole (Recruitment Closed); Arm C1: Palbociclib, trastuzumab and endocrine therapy; Arm C2: Treatment based of physician's choice
Drug: Chemotherapy — Gemcitabine, vinorelbine, capecitabine, eribulin or a taxane
  Other Names: CT
  Arms: Arm C2: Treatment based of physician's choice
Drug: Antibody-Drug Conjugates — 3.6 mg/kg iv every 3 weeks
  Other Names: Trastuzumab emtansine (TDM-1)
  Arms: Arm C2: Treatment based of physician's choice

SUMMARY:
PATRICIA is a phase II, open-label, multicentre, Simon's two-stage-design study of the combination of palbociclib plus trastuzumab, with or without letrozole, in post-menopausal patients with HER2-positive locally advanced or metastatic breast cancer (MBC) who have received chemotherapy and treatment with trastuzumab for their metastatic disease. Cohorts A, B1, and B2 based on their HR status and treatment allocation were planned.

Cohort A included patients with hormone receptor-negative, HER2 positive breast cancer, who received trastuzumab + palbociclib.

Cohort B1 included patients with hormone receptor-positive, HER2 positive breast cancer, who received trastuzumab + palbociclib.

Cohort B2 included patients with hormone receptor-positive, HER2 positive breast cancer, who received trastuzumab + palbociclib + letrozole.

The aim of the PATRICIA study is to test the hypothesis that the addition of Palbociclib to standard therapy is well tolerated and can provide a benefit in progression-free survival.

Based on interim results from this trial that support the benefit of CDK4 / 6 inhibition in luminal disease, two additional cohorts will be included.

DETAILED DESCRIPTION:
After the amendment of PATRICIA study, two additional cohorts will be included:

* Cohort C1: will include patients with OR+, HER2 positive, Luminal intrinsic subtype determined by PAM50 who will receive trastuzumab + palbociclib + endocrine therapy (ET)
* Cohort C2: will include patients with OR+, HER2 positive, Luminal intrinsic subtype determined by PAM50 who will receive treatment of physician's choice.

When the recruitment of those cohorts C begins, the recruitment in cohorts A and B will be closed.

For cohorts C, an adaptive design will be applied to compare arms of treatment in patients with Luminal subtype locally advanced or metastatic breast cancer (MBC).

All patients in those cohorts will have histologically- confirmed HR+/HER2-positive and PAM50-confirmed Luminal intrinsic subtype breast adenocarcinoma, and must have received at least 1 previous line of sistemic treatment for locally advanced disease or MBC which must have included trastuzumab and/or anti-HER2 Antibody-Drug conjugate.

Stratification factors will include number of previous regimens for advanced breast cancer (one and two vs three or more) and presence of visceral disease (yes vs no).

Treatment in all cohorts will be administered until progression, unacceptable toxicity, patient consent withdrawal, or death A total of 102 patients will be included. The inclusion period will be divided in two phases. During phase I it is planned to include 45 patients in 24 months; considering early stopping rule according to SF rate. During phase II, the trial will continue until the final evaluable number of 102 randomizations are included.

ELIGIBILITY:
Inclusion Criteria

For Cohorts A and B (Recruitment Closed)

1. Written signed Informed Consent for all study procedures in accordance with the local administrative requirements prior to starting the protocol-specific procedures.
2. Female patients
3. Age 18 years or older
4. ECOG performance status 0 or 1.
5. Invasive HER2 positive breast cancer, according to the local laboratory, defined according to ASCO/CAP criteria as:

   1. 3+ overexpression on immunohistochemistry (>10% of invasive tumor cells with intensive, circumferential membrane staining)
   2. Positive in situ hybridization (FISH/CISH/SISH) in >10% of invasive tumor cells, having counted at least 20 cells in the area and based on:

   i. Single-probe HER2 gene copy number ≥ 6 signals/cell. ii. Dual-probe HER2/CEP17 ratio ≥ 2.0 with a mean HER2 gene copy number ≥ 4.0 signals/cell; HER2/CEP17 ratio ≥ 2.0 and < 4.0 signals/cell; and HER2/CEP17 ratio < 2.0 and ≥ 6.0 signals/cell.
6. Known hormone receptor, determined locally according to ASCO/CAP guidelines; OR or PgR considered positive in case of ≥1% of cell nuclei positive.
7. Histologically-confirmed adenocarcinoma of the breast, metastatic or locally advanced.

   1. Patients with locally advanced disease must have recurrent or progressive disease unsuitable for resection with curative intent. Patients with standard curative options available will not be eligible.
   2. In patients with bilateral breast cancer, HER2+ positivity must be demonstrated in both sites or in a metastatic biopsy.
8. All patients must have received at least 2 (maximum 4) previous lines of systemic treatment for metastatic or locally advanced disease, at least one of which must have included trastuzumab. Previous use of other anti-HER2 treatment, alone or in combination with chemotherapy, is permitted, including lapatinib, neratinib, pertuzumab or T-DM1. Previous use of any chemotherapy or hormone agent is permitted.
9. Tumour tissue available for biomarker analysis, obtained from metastatic lesions (preferably) or from the primary tumor.
10. Measurable or non-measurable (but evaluable) disease according to RECIST v1.1 criteria. (Appendix 5).
11. Adequate organ function, defined as:

    1. Absolute neutrophil count (ANC) ≥ 1.5 x 109/L.
    2. Haemoglobin (Hb) ≥9 g/dl (transfusion or use of EPO is permitted).
    3. Platelets > 100,000/mm3.
    4. Creatinine ≤ 1.5 x normal value
    5. AST or ALT ≤ 2.5 x ULN (or ≤5 x ULN in case of liver metastasis).
    6. Alkaline phosphatase ≤2.5 x ULN. Alkaline phosphatase may be more than 2.5 x ULN only in the case of bone metastases, and AST and ALT less than 1.5 x ULN.
    7. Total bilirubin ≤1.5 mg/dl (higher bilirubin levels are permitted if the patient has Gilbert's syndrome).
12. Baseline LVEF ≥50% measured using echocardiogram or equilibrium isotopic ventriculography (MUGA).
13. Absence of psychological, family, sociological or geographical conditions that could potentially hinder compliance with the study protocol and follow-up schedule. These situations must be discussed with the patient before she is included in the study. ..14. Postmenopausal status defined as previous bilateral oophorectomy, age >60 or <60, and amenorrhoea for at least 12 months (in absence of chemotherapy, tamoxifen, toremifene or ovarian suppression) and FSH and estradiol in postmenopausal range, according to local laboratory.

For cohorts C:

1. Written signed Informed Consent for all study procedures in accordance with the local administrative requirements prior to starting the protocol-specific procedures.
2. Male or female patients. Premenopausal or postmenopausal women.
3. Age 18 years or older.
4. ECOG performance status 0 to 2.
5. Invasive HER2 positive breast cancer, according to the central laboratory, defined according to ASCO/CAP criteria.
6. Hormone receptor positive (HR+), determined locally according to ASCO/CAP guidelines; OR or PgR considered positive in case of ≥1% of cell nuclei positive.
7. Centrally confirmed Luminal intrinsic subtype as per PAM50 analysis (i.e. Luminal A or Luminal B).
8. Histologically confirmed adenocarcinoma of the breast, metastatic or locally advanced.

   1. Patients with locally advanced disease must have recurrent or progressive disease unsuitable for resection with curative intent. Patients with standard curative options available will not be eligible.
   2. In patients with bilateral breast cancer, HER2+ positivity must be demonstrated in both sites or in a metastatic biopsy.
9. All patients must have received at least 1 previous line of systemic treatment for metastatic or locally advanced disease, at least one of which must have included trastuzumab and/or anti-HER2 Antibody-Drug conjugate). Previous use of other anti-HER2 treatment, alone or in combination with chemotherapy, is permitted, including but not limited to lapatinib, neratinib, pertuzumab or T-DM1. Previous use of any chemotherapy or hormone agent is permitted. Also patients who recur during or within 12 months after completing adjuvant treatment with trastuzumab and/or antiHER2-ADCs (including but not limited to T-DM1) can be enrolled in the moment of the diagnosis of metastatic disease.
10. Tumour tissue available for biomarker analysis, obtained from metastatic lesions (preferably) or from the primary tumour.
11. Measurable or non-measurable (but evaluable) disease according to RECIST 1.1 criteria.
12. Adequate organ function, defined as:

    1. Absolute neutrophil count (ANC) ≥ 1.5 x 109/L.
    2. Hemoglobin (Hb) ≥9 g/dl (transfusion or use of EPO is permitted).
    3. Platelets > 100,000/mm3
    4. Creatinine ≤ 1.5 x normal value
    5. AST or ALT ≤ 2.5 x ULN (or ≤5 x ULN in case of liver metastasis)
    6. Alkaline phosphatase ≤2.5 x ULN. Alkaline phosphatase may be more than 2.5 x ULN only in the case of bone metastases, and AST and ALT less than 1.5 x ULN.
    7. Total bilirubin ≤1.5 mg/dl (higher bilirubin levels are permitted if the patient has Gilbert's syndrome).
13. Baseline LVEF ≥50% measured using echocardiogram or equilibrium isotopic ventriculography (MUGA).
14. Absence of psychological, family, sociological or geographical conditions that could potentially hinder compliance with the study protocol and follow-up schedule. These situations must be discussed with the patient before she is included in the study.
15. If female of childbearing potential, must have a negative result of serum pregnancy test performed within 7 days prior to the first dose of study treatment.
16. Participants with a history of treated CNS metastases are eligible, provided they meet all of the following criteria:

    * Disease outside the CNS is present.
    * No evidence of interim progression between the completion of CNS-directed therapy and the screening radiographic study.
    * No history of intracranial hemorrhage or spinal cord hemorrhage.
    * Stable doses or no need of corticosteroids and anti-convulsants for symptomatic control
    * Minimum of 3 weeks between completion of CNS radiotherapy and Cycle 1 Day 1 of study treatment; and recovery from any significant (Grade ≥ 3) acute toxicity

Exclusion criteria

For cohorts A, B (Recruitment Closed)

1. Treatment with any investigational anticancer drug within 14 days of the start of study treatment.
2. Patient has received more than 4 previous lines of treatment (anti-HER2 drug +/- chemotherapy) for metastatic breast cancer or locally advanced disease. Exclusively hormonal treatments will not be taken into account.
3. Previous treatment with a cyclin-dependent kinase inhibitor.
4. History of other malignant tumours in the past 5 years, with the exception of adequately treated in situ carcinoma of the cervix, non-melanoma carcinoma of the skin, uterine cancer in stage I or other malignant tumours with an expected curative outcome.
5. Radiation therapy for metastases outside the brain carried out in the 21 days prior to inclusion in the study and/or patients who have received radiation to > 30% of the bone marrow.
6. Symptomatic hypercalcemia requiring treatment with bisphosphonates in the 21 days prior to inclusion in the study. Biphosphonates will be permitted for the prevention of bone events.
7. History of exposure to cumulative anthracycline doses greater than follows:

   1. Adriamycin > 400 mg/m2
   2. Epirubicin > 720 mg/m2
   3. Mitoxantrone > 120 mg/m2
   4. Idarubicin > 90 mg/m2
   5. If another anthracycline or more than one anthracycline has been used, the cumulative dose must not exceed the equivalent of 400 mg/m2 of adriamycin.
8. Cardiopulmonary dysfunction, defined as:

   1. Uncontrolled hypertension (systolic > 150 mmHg and/or diastolic > 100 mmHg) despite optimum medical treatment.
   2. Angina pectoris or arrhythmia poorly controlled with optimum medical treatment.
   3. History of congestive heart failure NCI CTCAE version 4.0 grade ≥ 3 NYHA class ≥ 2.
   4. History of LVEF decrease to < 40% or symptomatic congestive heart failure during prior treatment with trastuzumab.
   5. Myocardial infarction within 6 months before randomisation.
   6. Resting dyspnoea due to complications of the malignant disease, requiring continuous oxygen therapy.
9. Any other severe, uncontrolled disease (pulmonary, cardiac, metabolic, or haematological disorder, wound healing disorders, ulcers, bone fractures, infectious processes).
10. Major surgery in the 28 days prior to randomisation or foreseeable during study treatment period.
11. Infection with HIV or active Hepatitis B and/or Hepatitis C.
12. History of trastuzumab intolerance, including grade 3-4 infusion reaction or hypersensitivity.
13. Known hypersensitivity to any of the study drugs, including inactive ingredients.
14. Inability, in the opinion of the investigator, to comply with the protocol requirements or any comorbidity that might hinder study follow-up, response evaluation or the informed consent process.

Exclusion criteria Cohort C

1. Treatment with any investigational anticancer drug within 14 days of the start of study treatment.
2. Previous treatment with a cyclin-dependent kinase inhibitor.
3. History of other malignant tumors in the past 3 years, with the exception of adequately treated in situ carcinoma of the cervix, non-melanoma carcinoma of the skin, uterine cancer in stage I or other malignant tumors with an expected curative outcome.
4. Radiation therapy for metastases outside the brain carried out in the 21 days prior to inclusion in the study and/or patients who have received radiation to > 30% of the bone marrow.
5. Symptomatic hypercalcemia requiring treatment with bisphosphonates in the 21 days prior to inclusion in the study. Bisphosphonates or RANKL inhibitors will be permitted for the prevention of bone events.
6. History of exposure to cumulative anthracycline doses greater than follows:

   1. Adriamycin > 400 mg/m2
   2. Epirubicin > 720 mg/m2
   3. Mitoxantrone > 120 mg/m2
   4. Idarubicin > 90 mg/m2
   5. If another anthracycline or more than one anthracycline has been used, the cumulative dose must not exceed the equivalent of 400 mg/m2 of adriamycin.
7. Cardiopulmonary dysfunction, defined as:

   1. Uncontrolled hypertension (systolic > 150 mmHg and/or diastolic > 100 mmHg) despite optimum medical treatment.
   2. Angina pectoris or arrhythmia poorly controlled with optimum medical treatment.
   3. History of congestive heart failure NCI CTCAE version 5.0 grade ≥ 3 NYHA class ≥ 2.
   4. History of LVEF decrease to < 40% or symptomatic congestive heart failure during prior treatment with trastuzumab.
   5. Myocardial infarction within 6 months before randomization.
   6. Resting dyspnea due to complications of the malignant disease, requiring continuous oxygen therapy.
8. Any other severe, uncontrolled disease (pulmonary, cardiac, metabolic, or hematological disorder, wound healing disorders, ulcers, bone fractures, infectious processes).
9. Major surgery in the 28 days prior to randomization or foreseeable during study treatment period.
10. Infection with HIV or active Hepatitis B and/or Hepatitis C.
11. History of trastuzumab intolerance, including grade 3-4 infusion reaction or hypersensitivity.
12. Known hypersensitivity to any of the study drugs, including inactive ingredients.
13. Inability, in the opinion of the investigator, to comply with the protocol requirements or any comorbidity that might hinder study follow-up, response evaluation or the informed consent process.

In cohort C, patients that are initially allocated in the control arm (physician's treatment choice) and have a documented disease progression can be re-randomized to receive the experimental or control treatment (if they meet the inclusion criteria after progression).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 73 (Actual)
Dates: Start 2015-07 (Actual); Primary Completion 2023-09-29 (Actual); Study Completion 2023-11-30 (Actual)

PRIMARY OUTCOMES:
Progression-Free Survival at 6 months | From randomization date to date of first documentation of progression or death , whichever came first, assessed up to 6 months.
  For cohorts A,B1 and B2: This was defined as the proportion of patients alive and without progression (according to RECIST v1.1 criteria), 6 months after randomization.
Progression-Free Survival (PFS)as Assessed by the Investigator [ Time Frame: From randomization date to date of first documentation of progression or death | From randomization date to date of first documentation of progression or death , whichever came first, assessed up to 4 years
  For cohorts C: This will be defined as the proportion of patients alive and without progression (according to RECIST v1.1 criteria)

SECONDARY OUTCOMES:
Rate of Disease control rate (DCR) in treatment arms (A and B) | up to 5 years
  Number of patients with objective response (complete or partial) or stable disease according to RECIST 1.1 criteria for at least 12 weeks.
Rate of Overall tumour objective response rate (ORR) in treatment arms (A and B). | up to 5 years
  Number of patients who achieve complete or partial response according to RECIST 1.1 criteria during treatment.
Evaluation of time to progression (Cohorts A and B) | up to 5 years
  Time between treatment start and disease progression
Cardiac Safety profile in arms A and B: Percentage of Participants with cardiac adverse events | up to 5 years
  Frequency of cardiac events of any grade, frequency of grade III-IV grade cardiac events according to NYHA classification.
Overall Survival in treatment arms (Cohorts A and B). | up to 5 years
  Measured as time between treatment start and all-cause death.
Rate of Disease control rate (DCR) in both treatment arms (C1 and C2) | up to 4 years
  Number of patients with objective response (complete or partial) or stable disease according to RECIST 1.1 criteria for at least 8 weeks.
Rate of Overall tumour objective response rate (ORR) in treatment arms (C1 and C2). | up to 4 years
  Number of patients who achieve complete or partial response according to RECIST 1.1 criteria during treatment.
Median duration of response in both treatment arms (C1 and C2). | up to 4 years
  Time of median duration of response according to RECIST 1.1 by treatment arm.
Change From Baseline Between Treatment Comparison in Functional Assessment of Cancer Therapy FACT-B to assess patient reported breast cancer specific health related quality of life (HRQOL) and general health status in both treatment arms (C1 and C2). | From the date of randomization up to 5 years
  The FACT-B consists of the Functional Assessment of Cancer Therapy-General (FACT-G) (27-items) and a breast-specific module: a 10-item instrument designed to assess patient concernsrelating to BC. The FACT-G is a 27-item compilation of general questions divided into 4 domains: Physical Well-Being, Social/Family Well-Being, Emotional Well-Being, and Functional Well-Being. Patients are asked to respond to a Likert scale where 0=not at all, 1=a little bit, 2=somewhat, 3=quite a bit, and 4=very much.
Change From Baseline Between Treatment Comparison in Euroqol-5D (EQ-5D) to assess patient reported breast cancer specific health related quality of life (HRQOL) and general health status in both treatment arms (C1 and C2). | From the date of randomization up to 5 years
  The EuroQol EQ-5D is designed to assess health status in terms of a single index value or utility score. It contains 5 descriptors of current health state (mobility, self-care, usual activities, pain or discomfort, and anxiety or depression) with each dimension having 5 levels of function (1=no problem, 2=slight problem, 3=moderate problem, 4=severe problem, and 5=unable/extreme). The scores on the 5 descriptors are summarized to create a single summary score. The EQ-5D also includes a visual analog scale (VAS), in which the patients self-rate their overall health status on a scale from 0 (worst imaginable) to 100 (best imaginable).
Safety profile in all treatment arms: Percentage of Participants with Adverse Events | up to 5 years
  Measurements used to assess the safety profile will include adverse events of any grade, grade 3 and 4 adverse events, withdrawals due to adverse events and dose reductions due to adverse events. CTCAE v.5.0 will be used to evaluate AE grade.
To investigate biomarkers as predictors of response or resistance to the study treatment. | up to 5 years
  Beyond PAM50 test, peripheral blood samples will be collected, and plasma extracted for circulating tumoral DNA (ctDNA) determination.

CONTACTS AND LOCATIONS:
Overall Officials: Eva Ciruelos, MD, Principal Investigator — SOLTI Breast Cancer Research Group
Locations (35):
- Spain (35):
  - ICO-Badalona, Badalona, Barcelona
  - Hospital General De Catalunya, Sant Cugat del Vallès, Barcelona
  - Hospital Universitario Rey Juan Carlos, Móstoles, Madrid
  - Complejo Hospitalario Universitario A Coruña, A Coruña
  - Hospital General Universitario de Alicante, Alicante
  - Hospital Universitario de Badajoz, Badajoz
  - Hospital Clínic de Barcelona, Barcelona
  - Hospital de la Santa Creu i Sant Pau, Barcelona
  - Hospital Universitario del Vall d' Hebron, Barcelona
  - ICO Hospitalet, Barcelona
  - Hospital de Basurto, Bilbao
  - Consorcio Hospitalario Provincial de Castellón, Castellon
  - Hospital San Pedro de Alcantara, Cáceres
  - Hospital Reina Sofía de Córdoba, Córdoba
  - Hospital Universitario Virgen de las Nieves, Granada
  - HU Clínico San Cecilio, Granada
  - Complejo Asistencial Universitario de León, León
  - HU Arnau de Vilanova Lleida, Lleida
  - Centro Integral Oncológico Clara Campal (CIOCC), Madrid
  - H. Severo Ochoa, Madrid
  - H. U Puerta de Hierro, Madrid
  - Hospital Universitario Doce de Octubre, Madrid
  - Hospital Universitario Ramon y Cajal, Madrid
  - Hospital Son Llatzer, Palma de Mallorca
  - Hospital Universitario Son Espases, Palma de Mallorca
  - Complejo Hospitalario de Navarra, Pamplona
  - Hospital Universitario de Salamanca, Salamanca
  - Hospital Virgen Universitario Virgen de Macarena, Seville
  - Hospital Quirón Salud Sagrado Corazón, Seville
  - Hospital Universitario Virgen del Rocio, Seville
  - Hospital Universitario Sant Joan de Reus, Tarragona
  - Instituto Valenciano de Oncología, Valencia
  - Hospital General Universitario de Valencia, Valencia
  - Hospital Clinico Universitario de Valencia, Valencia
  - Hospital Álvaro Cunqueiro, Vigo

REFERENCES:
- [Background] Ciruelos E, Villagrasa P, Pascual T, Oliveira M, Pernas S, Pare L, Escriva-de-Romani S, Manso L, Adamo B, Martinez E, Cortes J, Vazquez S, Perello A, Garau I, Mele M, Martinez N, Montano A, Bermejo B, Morales S, Echarri MJ, Vega E, Gonzalez-Farre B, Martinez D, Galvan P, Canes J, Nuciforo P, Gonzalez X, Prat A. Palbociclib and Trastuzumab in HER2-Positive Advanced Breast Cancer: Results from the Phase II SOLTI-1303 PATRICIA Trial. Clin Cancer Res. 2020 Nov 15;26(22):5820-5829. doi: 10.1158/1078-0432.CCR-20-0844. Epub 2020 Sep 16. PMID 32938620
- [Derived] Peddi PF, Slamon DJ. Frontiers in HER2-positive breast cancer in 2020. Curr Opin Obstet Gynecol. 2021 Feb 1;33(1):48-52. doi: 10.1097/GCO.0000000000000677. PMID 33369581